CLINICAL TRIAL: NCT00371033
Title: A Randomized, Placebo-controlled Multi-center Clinical Trial to Evaluate the Efficacy and Safety of Pregabalin for the Treatment of Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS)
Brief Title: Efficacy & Safety Study of Pregabalin to Treat Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS)
Acronym: CPCRN RCT#2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CPCRN2 Pregabalin; U01DK065209 (NIH)
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS)
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pregabalin (Active Comparator)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 150 mg/d (50 mg orally 3 times daily) for 2 weeks, then 300 mg/d (100 mg orally 3 times daily) for 2 weeks, and then 600 mg/d (200 mg orally 3 times daily) for 2 weeks.
  Arms: Pregabalin
Drug: Placebo — Placebo at same frequency as pregabablin
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether pregabalin is an effective treatment for Chronic Prostatitis/Chronic Pelvic Pain Syndrome.

DETAILED DESCRIPTION:
Primary Objectives

1. To compare six (6) weeks of treatment with pregabalin versus placebo in CP/CPPS participants with respect to the primary endpoint in the NIH-CPSI
2. To evaluate the safety and tolerability of six (6) weeks of pregabalin in CP/CPPS participants

Design

Eligible participants will receive either pregabalin or placebo, randomly assigned at a ratio of 2:1. Study treatment will be for 6 weeks with dose starting at 150mg going up to 300mg and finally to 600mg daily, to maximum tolerated dose. Participants will be advised to take the study medication 3 times per day. There are 3 clinic visits and 2 telephone contacts. Participants will be offered optional active treatment for an additional 6 weeks at the end of the first 6 weeks. For those participating in both phases there are a total of 4 clinic visits and 5 telephone contacts.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed and dated the appropriate Informed Consent document.
* Participant must have had symptoms of discomfort or pain in the pelvic region for at least a three (3) month period within the last six (6) months.

Exclusion Criteria:

* Participant has continued evidence of facultative Gram negative or enterococcus with a value of ≥ 1000 and ≤ 100,000 CFU/ml in mid-stream urine (VB2), as demonstrated by repeat culture obtained no less than seven (7) days post antibiotic treatment.
* Participant has a calculated creatinine clearance of <60 mL/min.
* Participant has a platelet count <100,000/mm3.
* Participant is allergic to antiepileptic/antiseizure medications.
* Participant has a known allergy or sensitivity to pregabalin (Lyrica®).
* Participant is taking thiazolidinedione antidiabetic agents (i.e. rosiglitazone and pioglitazone).
* Participant has New York Heart Association Class III or IV congestive heart failure.
* Participant has a history of thrombocytopenia, or a bleeding diathesis.
* Participant has a history of prostate, bladder or urethral cancer.
* Participant has a history of alcohol abuse.
* Participant has inflammatory bowel disease (such as Crohn's disease or ulcerative colitis, but not irritable bowel syndrome).
* Participant has undergone pelvic radiation or systemic chemotherapy.
* Participant has undergone intravesical chemotherapy.
* Participant has been treated with intravesical BCG.
* Participant has unilateral orchalgia without other pelvic symptoms.
* Participant has an active urethral stricture.
* Participant has a neurological disease or disorder affecting the bladder.
* Participant has a neurological impairment or psychiatric disorder preventing his understanding of consent and his ability to comply with the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kusek, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Lee Nyberg, PhD, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (11):
- United States (10):
  - Charles R Drew University of Medicine & Science, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Harvard Medical School, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - University of Washington Harborview Medical Center, Seattle, Washington
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/cpcrn2-rct2/?query=cpcrn2
URL: https://repository.niddk.nih.gov/studies/cpcrn2-rct2/?query=cpcrn2

REFERENCES:
- [Derived] Pontari MA, Krieger JN, Litwin MS, White PC, Anderson RU, McNaughton-Collins M, Nickel JC, Shoskes DA, Alexander RB, O'Leary M, Zeitlin S, Chuai S, Landis JR, Cen L, Propert KJ, Kusek JW, Nyberg LM Jr, Schaeffer AJ; Chronic Prostatitis Collaborative Research Network-2. Pregabalin for the treatment of men with chronic prostatitis/chronic pelvic pain syndrome: a randomized controlled trial. Arch Intern Med. 2010 Sep 27;170(17):1586-93. doi: 10.1001/archinternmed.2010.319. PMID 20876412

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-Pregabalin: Men were randomly assigned to receive pregabalin or placebo in a 2:1 ratio and were treated for 6 weeks. Treatment dosage was escalated as follows: 150 mg/d (50 mg orally 3 times daily) for 2 weeks, then 300 mg/d (100 mg orally 3 times daily) for 2 weeks, and then 600 mg/d (200 mg orally 3 times daily) for 2 weeks. Men assigned to receive placebo underwent a similar escalation in the number of capsules prescribed.
- 2-Placebo: Men were randomly assigned to receive pregabalin or an identical placebo in a 2:1 ratio and were treated for 6 weeks. Treatment dosage was escalated as follows: 150 mg/d (50 mg orally 3 times daily) for 2 weeks, then 300 mg/d (100 mg orally 3 times daily) for 2 weeks, and then 600 mg/d (200 mg orally 3 times daily) for 2 weeks. Men assigned to receive placebo underwent a similar escalation in the number of capsules prescribed.
Period: Overall Study
Arm/Group | 1-Pregabalin | 2-Placebo
Started | 218 | 106
Completed | 210 | 103
Not Completed | 8 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — No longer interested | 2 | 0
Not completed — Uknown | 3 | 1

BASELINE CHARACTERISTICS:
Population: Based on evaluable participants
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Pregabalin | 2-Placebo | Total
Number analyzed (Participants) | 216 | 103 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (13.0) | 45.2 (12.2) | 47.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 216 | 103 | 319
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 24 | 14 | 38
  White | 178 | 75 | 253
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 11 | 2 | 13
NIH-CPSI total score (possible score, 0-43) [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI) measures the 3 key domains of Chronic Prostatitis/Chronic Pelvic Pain Syndrome: pain (location, frequency, and severity; possible score, 0-21), urinary symptoms (irritative and obstructive; possible score, 0-10), and impact/quality of life (possible score, 0-12), for a total possible score of 0 to 43. A higher score indicates more severe symptoms.
  units on a scale | 26.2 (5.6) | 25.9 (6.1) | 26.1 (5.7)
NIH-CPSI pain subscore (possible score, 0-21) [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI) pain subscore is determined by location, frequency, and severity of pain symptoms with a possible score of 0-21. A higher score indicates more severe symptoms.
  units on a scale | 12.3 (3.0) | 12.4 (3.1) | 12.4 (3.0)
NIH-CPSI urinary symptoms subscore (possible score, 0-10) [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI) urinary subscore measures irritative and obstructive symptoms with a possible score of 0-10. A higher score indicates more severe symptoms.
  units on a scale | 4.9 (2.7) | 4.7 (2.7) | 4.8 (2.7)
NIH-CPSI QOL subscore (possible score, 0-12) [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI) impact/quality of life subscore measures participant-reported symptoms with a possible score, 0-12. A higher score indicates more severe symptoms.
  units on a scale | 8.9 (2.0) | 8.9 (2.0) | 8.9 (2.0)
SF-12 PCS score (possible score, 0-100) [Mean (Standard Deviation); unit: units on a scale] — The Medical Outcomes Study 12-item Short Form Survey (SF-12) is a general health questionnaire that is comprised of a mental component score (MCS-12) and a physical component score (PCS-12). The SF-12 ranges from 0-100 for the Physical [PCS] and Mental [MCS] Component Summary scores, with the mean set at 50 and higher scores indicating better quality of life. Population: Based on evaluable patient data
  units on a scale
    number analyzed (Participants) | 213 | 102 | 315
    (all) | 44.9 (10.1) | 43.9 (10.3) | 44.6 (10.2)
SF-12 MCS score (possible score, 0-100) [Mean (Standard Deviation); unit: units on a scale] — The Medical Outcomes Study 12-item Short Form Survey (SF-12) is a general health questionnaire that is comprised of a mental component score (MCS-12) and a physical component score (PCS-12). The SF-12 ranges from 0-100 for the Physical [PCS] and Mental [MCS] Component Summary scores, with the mean set at 50 and higher scores indicating better quality of life. Population: Based on evaluable patient data
  units on a scale
    number analyzed (Participants) | 213 | 102 | 315
    (all) | 41.8 (10.6) | 42.8 (10.6) | 42.1 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Decrease in the NIH-CPSI Total Score by at Least 6 Points
Description: Decrease (improvement) in the National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI) score of at least 6 points from baseline to week 6. The NIH-CPSI measures the 3 key domains of CP/CPPS: pain (location, frequency, and severity; possible score, 0-21), urinary symptoms (irritative and obstructive; possible score, 0-10), and impact/quality of life (possible score, 0-12), for a total possible score of 0 to 43. A 6-point decrease in NIHCPSI score has been shown to be clinically perceptible in previous clinical trials of men with CP/CPPS.
Time Frame: Baseline and 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 1-Pregabalin: Randomized to Pregabalin
- 2-Placebo: Randomized to placebo
Arm/Group | 1-Pregabalin | 2-Placebo
Number analyzed (Participants) | 218 | 106
Participants | 103 | 38

2. Secondary Outcome: Subscales of the NIH-CPSI
Description: The National Institutes of Health -Chronic Prostatitis Symptom Index (NIH-CPSI) measures the 3 key domains of Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS): pain (location, frequency, and severity; possible score, 0-21), urinary symptoms (irritative and obstructive; possible score, 0-10), and impact/quality of life (possible score, 0-12), for a total possible score of 0 to 43. A higher score indicates more severe symptoms. A 6-point decrease in NIHCPSI score has been shown to be clinically perceptible in previous clinical trials of men with CP/CPPS.
Time Frame: 6 weeks
Population: The overall number of participants analyzed in the secondary outcome measures were 210 for the pregabalin arm and 103 for the placebo arm.
Measure: Mean (Standard Deviation); unit: units on the NIH-CPSI scale
Arm/Group | 1-Pregabalin | 2-Placebo
Number analyzed (Participants) | 210 | 103
units on the NIH-CPSI scale
  Total score | 19.7 (8.5) | 21.6 (8.9)
  Pain domain score | 9.1 (3.1) | 10.1 (4.7)
  Urinary symptoms domain score | 3.7 (2.6) | 4.0 (2.7)
  Quality of life domain | 6.9 (2.9) | 7.4 (3.1)

3. Secondary Outcome: Moderately or Markedly Improve on Global Response Assessment (GRA)
Description: The GRA is a 7-question patient self-reported assessment that measures perception of change in symptoms (improvement, no change, or deterioration). The responses are centered at zero (no change in symptoms). Men who reported that they were moderately or markedly improved on a 7-point GRA at the end of the study were identified as treatment responders.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Pregabalin | 2-Placebo
Number analyzed (Participants) | 218 | 106
Participants | 68 | 20

4. Secondary Outcome: Hospital Anxiety & Depression Scale
Description: Hospital Anxiety and Depression Scale (HADS) (range, 0-42, with higher scores indicating greater anxiety and depression)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1-Pregabalin | 2-Placebo
Number analyzed (Participants) | 210 | 103
units on a scale | 12.4 (7.8) | 12.2 (7.8)

5. Secondary Outcome: McGill Pain Questionnaire
Description: The McGill Pain Questionnaire (MPQ) evaluates the quality of pain as well as the intensity of pain. The McGill Pain Questionnaire ranges from 0-45 for a total pain score, and is the sum of a sensory subscore of 0-33 and affective subscore of 0-12. Higher scores indicate greater pain.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1-Pregabalin | 2-Placebo
Number analyzed (Participants) | 210 | 103
units on a scale | 9.6 (8.8) | 12.4 (9.1)

6. Secondary Outcome: Medical Outcomes Study Short Form 12
Description: Medical Outcomes Study 12-Item Short Form Health Survey (SF-12) (range, 0-100 for the Physical [PCS] and Mental [MCS] Component Summary scores, with the mean set at 50 and higher scores indicating better quality of life)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1-Pregabalin | 2-Placebo
Number analyzed (Participants) | 210 | 103
units on a scale
  Physical [PCS] Component Summary | 46.9 (10.1) | 44.3 (10.6)
  Mental [MCS] Component Summary | 45.0 (11.2) | 44.6 (10.6)

7. Secondary Outcome: Sexual Health Inventory for Men
Description: Sexual Health Inventory for Men (SHIM) (range, 1-25, with higher scores indicating better sexual function)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1-Pregabalin | 2-Placebo
Number analyzed (Participants) | 210 | 103
units on a scale | 16.4 (8.4) | 17.2 (7.8)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Final Adverse Events were reported by arm. They included all AEs by type, regardless of their relationship to study drug.
  Patients are counted once in each category and included in the column relating to their worst toxicity grade. Patients may have had events in more than one body system category. An adverse event is not counted if the same event is observed at baseline with an equal or greater toxicity grade.
Arm/Group | 1-Pregabalin | 2-Placebo
All-Cause Mortality (participants affected / at risk) | 0/218 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/218 | 0/106
Other Adverse Events (participants affected / at risk) | 129/218 | 62/106
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Pregabalin (N=218) | 2-Placebo (N=106)
Pain (General disorders) | 38 (38) | 35 (38) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Constitutional symptoms (General disorders) | 53 (53) | 22 (22) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Neurologic symptoms (Nervous system disorders) | 40 (40) | 20 (20) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Gastrointestinal disturbance (Gastrointestinal disorders) | 40 (40) | 20 (20) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Ocular/visual symptoms (Eye disorders) | 15 (15) | 3 (3) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Renal/genitourinary symptoms (Renal and urinary disorders) | 12 (12) | 2 (2) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No